CLINICAL TRIAL: NCT05332951
Title: Study of Empathy in Patients With Multiple Sclerosis
Brief Title: Study of Empathy in MS
Acronym: SEmPathy
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220241; 2022-A00713-40 (Other: IDRCB)
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis
Keywords: MS; social cognition; empathy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients followed for multiple sclerosis
  Interventions: Other: Interpersonal Reactivity Index

INTERVENTIONS:
Other: Interpersonal Reactivity Index — Questionnaire to be completed by the patient

SUMMARY:
Multiple sclerosis is a chronic inflammatory disease of the central nervous system whose exact etiology remains unclear, underpinned by multiple pathophysiological mechanisms, and is a cause of significant motor and cognitive disability.

Some studies report a prevalence of 40% to 60% of cognitive impairment during the disease, and represents a major factor influencing quality of life in patients with MS.

Cognitive impairment can affect one or more of the 6 cognitive functions, including social cognition and its three components: theory of mind, or an individual's ability to infer intention and other's behavior, empathy, and social perceptions and knowledge.

To date, few studies have focused on the more specific study of empathy in MS. They seem to suggest the existence of a deficit but rely on small numbers of patients.

There appear to be many confounding factors but their direct relationship to empathy is not clearly established: potentially related comorbidities, such as anxiety and depression that are frequently found in MS patients ; level of education and cognitive reserve; and finally the very characteristics of the disease.

Indeed, data concerning relationship between empathy and the activity or stage of MS seem so far contradictory.

Alexithymia, or inability to express feelings verbally, is a pathology close to empathy deficit, and can affect patients' daily lives in a similar way. Prevalence of alexithymia in MS patients has been shown to be higher than in general population, and its parallel study with empathy seems relevant.

The aim of this study is to assess the level of empathy on a larger scale of MS population and to study various confounding factors known to influence the level of empathy, such as anxiety, depression, level of education but also the characteristics of the disease: its duration of evolution, its stage, its activity, and associated disability.

The investigator team will conduct a prospective observational study in MS patients to assess their level of empathy versus a control population of healthy subjects and study the influence of these different variables.

DETAILED DESCRIPTION:
Multiple sclerosis is a chronic inflammatory disease of the central nervous system that affects more than 2.8 million people worldwide and whose diagnosis is most often made around the age of 30. Its prevalence is increasing since the 90s and seems to involve certain susceptibility genes and environmental factors.

This inflammatory disease, whose exact etiology remains unclear, underpinned by multiple pathophysiological mechanisms, is the cause of significant motor and cognitive disability. Indeed, some studies report a prevalence of 40% to 60% of cognitive impairment during the disease, and represents a major factor influencing quality of life in patients with MS.

Defined as a part of cognitive functions, social cognition refers to a set of processes involved in social interactions, including perception, understanding and reasoning about emotions and behaviors of others.

There are usually several components described within social cognition: - theory of mind, or an individual's ability to infer other's intention and behavior, - empathy, which is the ability to react to and understand other's emotion, and - social perceptions and knowledge (from prosody, bodily gestures and facial expressions).

The concept of empathy was first defined in the 19th century by Theodor Lipps, then one of the main representatives of German psychology, under the term "Einfühlung" as a tool for understanding the mental status of the other.

Several works have tried to distinguish between affective and cognitive empathy.

Affective empathy is defined as the affective state produced in response to emotional experiences of others. Cognitive empathy represents the understanding of an external situation from the point of view of the person who lives it by distinguishing the other from oneself. This last component is substantially related to the definition of theory of mind.

Empathy can be assessed via a 28-item IRI (Interpersonal Reactivity Index) self-questionnaire, the most commonly used test in clinical research, the French version of which has been validated on 322 subjects.

To date, few studies have focused on the more specific study of empathy in MS and its two aforementioned components but seem to suggest the existence of a deficit.

There appears to be many confounding factors but their direct relationship to empathy is not clearly established: potentially related comorbidities, such as anxiety and depression that are frequently found in MS patients ; level of education and cognitive reserve; and finally the very characteristics of the disease.

Indeed, data concerning relationship between empathy and the activity or stage of MS seem so far contradictory.

Alexithymia, or inability to express feelings verbally, is a pathology close to empathy deficit, and can affect patients' daily lives in a similar way. Prevalence of alexithymia in MS patients has been shown to be higher than in general population, and its parallel study with empathy seems relevant.

The aim of this study is to assess the level of empathy on a larger scale of MS population and to study various confounding factors known to influence the level of empathy, such as anxiety, depression, level of education but also the characteristics of the disease: its duration of evolution, its stage, its activity, and associated disability.

The investigator team conducted a prospective observational study in MS patients to assess their level of empathy versus a control population of healthy subjects and study the influence of these different variables.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 60
* Follow-up for multiple sclerosis meeting the revised McDonalds diagnostic criteria of 2017.
* Patient not objecting to participation in the research.

Exclusion Criteria:

NA

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients followed for multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Interpersonal Reactivity Index (IRI) | 5 minutes
  QUestionnaire IRI will be completed by patients

SECONDARY OUTCOMES:
alexithymia | 5 minutes
  Toronto Alexithymia Scale TAS 20 (rated from 20 to 100)
anxiety and depression | 5 minutes
  Hospital Anxiety and Depression Scale HADS will be completed by patients (rated from 0 to 21)
cognitive reserve | 5 minutes
  Cognitive Reserve Index questionnaire CRIq will be completed by patients
fatigue | 5 minutes
  Fatigue Severity Scale (FSS) will be completed by patients (rated from 9 to 63)
cognitive deficit | 3 minutes
  Symbol Digit Modalities Test (SDMT, rated from 0 to 90) to be defined by the investigator

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital de la Pitié Salpêtrière, Paris
  - Hôpital Saint Antoine, Paris